CLINICAL TRIAL: NCT02806180
Title: Single v Dual-Operator Ultrasound Technique for Peripheral Vascular Access in the Emergency Department
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Dr. Jordan Chenkin, Dr., Sunnybrook Health Sciences Centre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 410001002
Record Dates: First submitted 2016-06-15; First posted 2016-06-20 (Estimated); Last update posted 2016-06-20 (Estimated); Status verified 2016-06

CONDITIONS: Patients With Difficult Vascular Access.

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Single-Operator (Experimental): For the 'Single Operator Ultrasound Guided IV placement' arm the RN operator will use the ultrasound probe to identify the target vein, and continue to hold and adjust the probe while placing the IV.
  Interventions: Procedure: Single Operator Ultrasound Guided IV placement
- Dual-Operator (Experimental): For the 'Dual Operator Ultrasound Guided IV placement' arm the RN operator will use the US to identify the target vein, at which time the study coordinator will hold the ultrasound probe in position. The RN operator will then place the IV.
  Interventions: Procedure: Dual Operator Ultrasound Guided IV placement

INTERVENTIONS:
Procedure: Dual Operator Ultrasound Guided IV placement — Second operator holds ultrasound probe.
  Arms: Dual-Operator
Procedure: Single Operator Ultrasound Guided IV placement — Single operator holds ultrasound probe and places IV.
  Arms: Single-Operator

SUMMARY:
This is a randomized controlled trial comparing the success of US guided peripheral IV placement between single vs dual-operator technique among a convenience sample of patients with moderate or difficult vascular access in a tertiary care Emergency Department.

DETAILED DESCRIPTION:
Gaining intravenous (IV) access is a common and important procedure in the emergency department (ED). IV access is needed to deliver drugs, enable fluid resuscitation and sample blood, and delays in gaining access can lead to patient harm. Ultrasound (US) is a commonly used tool in the ED, and the utility of ultrasound in the placement of IVs in patients with difficult access has been well described. This study aims to further guide the use of this evidence based tool by ED Registered Nurses. The focus will be comparing single-operator technique, in which the same provider manipulates the ultrasound probe while simultaneously placing the IV, to a dual-operator technique whereby a second provider manipulates the probe. Any measured advantage has implications in guiding education and practice, as well as informing future ED policy.

ELIGIBILITY:
Inclusion Criteria:

* Adult (18 years and older) patients predicted to require intravenous cannulas and identified at triage as having moderate or difficult access based on the following criteria:

Moderate: peripheral vein is visible or palpable but difficulty is expected based on patient characteristics both clinical and historical.

Difficult: No peripheral veins visible or palpable, or two failed attempts by traditional landmarking (LM).

Exclusion Criteria:

* Exclusion criteria will include patients who have already undergone successful pre-hospital IV placement, patients with an indwelling vascular device, patients who are critically ill (Canadian Triage Acuity Score I) or objection to study enrolment by the attending MD for any reason. If no suitable target vein can be identified with US the patient data will be collected and the patient will be excluded from the statistical analysis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2016-07; Primary Completion 2017-07 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
First Pass Success | Total procedure time (<15 minutes)
  The proportion of patients in whom vascular access is obtained on the first attempt with a single skin puncture.

SECONDARY OUTCOMES:
Overall Success | Total procedure time (<15 minutes)
  The proportion of patients in whom vascular access is achieved within a maximum of three attempts at US guided placement.
Number of Attempts | Total procedure time (<15 minutes)
  Total number of individual skin punctures that a patient receives.
Time to Canulation | Total procedure time (<15 minutes)
  Measured as the time from when the Registered Nurse operator first picks up the ultrasound probe to the time when 'flashback' is seen to confirm placement.
Patient Pain Score | Total procedure time (<15 minutes)
  To be completed by the patient immediately after the procedure: 10cm visual analogue scale from 'painless' to 'very painful'.
Operator Ease of Use Score | Total procedure time (<15 minutes)
  To be completed by the Registered Nurse operator immediately after the procedure: 10cm visual analogue scale from 'very easy' to 'very difficult'.

CONTACTS AND LOCATIONS:
Overall Officials: Jordan Chenkin, MD, FRCPC, Principal Investigator — Sunnyrbook Health Science Centre, University of Toronto

IPD SHARING:
Plan to Share IPD: No